CLINICAL TRIAL: NCT04213937
Title: The Efficacy and Safety of Nab-paclitaxel Versus Topotecan As Second-Line Treatment for Patients With Extensive Stage Small Cell Lung Cancer: A Multicenter, Randomized Controlled Study
Brief Title: Nab-paclitaxel Versus Topotecan As Second-Line Treatment for Patients With Extensive Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jie Wang, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAL-SCLC-01
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: nab-paclitaxel Topotecan
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Topotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nab-paclitaxel (Experimental): nab-paclitaxel 125mg/m2, i.v. d1, d8, Repeated every 3 weeks for 4-6 cycles
  Interventions: Drug: nab-paclitaxel
- Topotecan (Active Comparator): Topotecan 1.25mg/m2/d, i.v, 1hour, d1-d5, Repeated every 3 weeks for 4-6 cycles.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: nab-paclitaxel — Drug: nab-paclitaxel 125mg/m2, i.v. d1, d8, Repeated every 3 weeks for 4-6 cycles.
  Arms: nab-paclitaxel
Drug: Topotecan — Drug: Topotecan 1.25mg/m2/d, i.v, 1hour, d1-d5, Repeated every 3 weeks for 4-6 cycles.
  Arms: Topotecan

SUMMARY:
The purpose of this study is to compare the efficacy and safety of nab-paclitaxel with topotecan as second-line treatment for patients with extensive stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 75years, male or female; 2.Histological or pathological diagnosis of small cell lung caner; 3.Progression or relapse after first-line chemotherapy, extensive disease; 4.ECOG performance status of 0-2; 5.Life expectancy of 3 months or more; 6.Patient must be accessible for treatment and follow-up; 7.For women of child-bearing age, the pregnancy test results (serum or urine) within 72 hours before enrolment must be negative. They will take appropriate methods for contraception during the study; 8.Signed informed consent.

Exclusion Criteria:

1. symptomatic brain metastases;
2. Uncontrolled serious medical conditions that, in the opinion of the investigator, would affect the ability of the subject to receive the study regimen, such as concomitant serious medical conditions, including severe heart disease, cerebrovascular disease, uncontrolled diabetes mellitus, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc.;
3. Have dementia, altered mental state or any mental illness that would prevent understanding or informed consent or fill out questionnaires;
4. Received any investigational drug within 30 days of the planned first dose of this study treatment.
5. Prior Grade ≥ 2 peripheral neuropathy(according to (NCI CTCAE), version 5.0);
6. Known to be hypersensitive, highly sensitive, or intolerant to study-related medications or their excipients;
7. Have malignant tumors in the past 5 years, except for clinically cured basal cell or squamous cell skin cancer, local prostate cancer after radical operation, and ductal carcinoma in situ after radical operation;
8. Bone marrow function: Neutrophils < 1.5×109/L, platelets < 100×109/L, hemoglobin < 90 g/L; Hepatic and renal function: Serum creatinine > 1.5×ULN; AST and ALT > 2.5×ULN or > 5×ULN in the presence of hepatic metastasis; Total bilirubin >1.5×ULN;
9. Patients need other anti-tumor drugs;
10. Known HIV, hepatitis B/C virus positive ;
11. The researchers considered the patients who were not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2020-01-31 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 1 years post treatment
  OS was defined as the time from the date of the first administration of trial regimen to the date of death from any cause (event) or last follow-up (censored data).

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1 years
  Response evaluation disease progression defined by Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1) criteria.
  Response (PR), refers to the number of cases with complete and partial response after treatment as a percentage of the total number of evaluable cases.
Progression free survival (PFS) | 1 years
  The time from treatment to tumor progression or death
Adverse events (AE) | 3 years
  Adverse events (AE) were monitored on an ongoing basis and classified according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0. Patients were assessed for toxicities before each administration, and toxicity was graded accordingly

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided